CLINICAL TRIAL: NCT03379506
Title: A Phase IIb Clinical Study to Assess the Pharmacokinetics, Safety, and Efficacy of the Combination Regimen of Elbasvir (EBR)/Grazoprevir (GZR) in Participants Aged 3 to Less Than 18 Years With Chronic Hepatitis C Infection
Brief Title: Elbasvir (EBR)/Grazoprevir (GZR) in Pediatric Participants With Chronic Hepatitis C Infection (MK-5172-079)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5172-079; MK-5172-079 (Other: Merck Protocol Number); 2015-003006-16 (EudraCT Number)
Record Dates: First submitted 2017-12-13; First posted 2017-12-20 (Actual); Results first posted 2020-08-17 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination; grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EBR/GZR (Experimental): Pediatric participants receive EBR/GZR as either FDC tablets or oral granules once daily for 12 weeks. A 24-week follow-up period will follow the 12-week treatment regimen.
  Interventions: Drug: EBR/GZR FDC Tablet; Drug: Placebo; Drug: Grazoprevir Oral Granules; Drug: Elbasvir Oral Granules

INTERVENTIONS:
Drug: EBR/GZR FDC Tablet — Participants who are 12 to <18 years of age will receive oral FDC tablets with EBR 50 mg/GZR 100 mg once daily by mouth.
  Other Names: MK-5172A; ZEPATIER®
Drug: Placebo — Placebo tablet matched to EBR/GZR FDC tablet.
Drug: Grazoprevir Oral Granules — Participants 3 to <12 years of age take grazoprevir granules 0.5 mg by mouth in a soft food vehicle at a dose not to exceed 50 mg.
  Other Names: MK-5172
Drug: Elbasvir Oral Granules — Participants 3 to <12 years of age take elbasvir oral granules 1 mg by mouth in a soft food vehicle at a dose not to exceed 100 mg.
  Other Names: MK-8742

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK), safety, and efficacy of oral MK-5172 (a fixed dose combination [FDC] tablet containing elbasvir [EBR] 50 mg and grazoprevir [GZR] 100 mg) and EBR/GZR (varying doses) pediatric granules in pediatric hepatitis C virus (HCV)-infected participants who are 3 to <18 years of age. Within each age cohort (Cohort 1: 12 to <18 years of age; Cohort 2: 7 to <12 years of age; and Cohort 3: 3 to <7 years of age), a Mini Cohort of 7 participants will be enrolled first. For the oldest cohort (Cohort 1), the Mini Cohort will assess ability to swallow a placebo tablet prior to administering active FDC tablets; participants in Cohorts 2 and 3 will take pediatric granules instead of a tablet.

ELIGIBILITY:
Inclusion Criteria:

* Has documented chronic HCV genotype (GT) 1 or GT4 infection
* Has the following liver disease staging assessment: absence of cirrhosis or compensated cirrhosis
* Has one of the following HCV treatment statuses:
* GT1 and GT4: treatment-naïve (TN), defined as no prior exposure to any interferon (IFN)-containing regimen, ribavirin (RBV), or other HCV-specific direct acting antiviral (DAA) agent
* GT1 only: treatment-experienced (TE) with no previous treatment with HCV specific DAA agents.
* If female is not pregnant, not breastfeeding, and is either not of childbearing potential or follows the contraceptive guidance during the treatment period and for at least 14 days after the last dose of study treatment.

Exclusion Criteria:

* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy, or other signs or symptoms of advanced liver disease.
* Is cirrhotic AND has a Child-Turcotte-Pugh score >6, corresponding to a Child Class B or C.
* Is co-infected with Human Immunodeficiency Virus (HIV).
* Has evidence of past or present hepatitis B infection.
* Has a history of malignancy ≤5 years prior to signing informed consent or is under evaluation for other active or suspected malignancy.
* Female expects to conceive or donate eggs from Day 1 through at least 14 days after the last dose of study treatment or longer.
* Has any of the following conditions: organ transplants other than cornea and hair; poor venous access; history of gastric surgery or malabsorption disorders; any clinically significant cardiac abnormalities/dysfunction that may interfere with participant treatment, assessment, or compliance; any major medical condition which might interfere with participant treatment, assessment, or compliance; history of a medical/surgical condition that resulted in hospitalization within the 3 months prior to enrollment; medical/surgical conditions that may result in a need for hospitalization during the study duration; any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, tumor necrosis factor antagonists, or immunosuppressant drugs; life-threatening serious adverse event (SAE) during the screening period; history of chronic hepatitis not caused by HCV.
* If female has a positive urine pregnancy test within 24 hours before the first dose of study treatment.
* Is taking or plans to take prohibited medications, or is taking herbal supplements.
* Has had previous HCV direct acting antiviral (DAA) treatment.
* Is currently participating or has participated in a study with an investigational compound within prior 30 days
* Has significant emotional problems or a clinically significant psychiatric disorder that may interfere with participant treatment, assessment, or compliance with the protocol.
* Has clinically relevant drug or alcohol abuse within prior 12 months that may interfere with participant treatment, assessment, or compliance.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (15):
- United States (8):
  - University of California San Francisco ( Site 0020), San Francisco, California
  - Florida Hospital ( Site 0006), Orlando, Florida
  - Children's Center for Advanced Pediatrics ( Site 0204), Atlanta, Georgia
  - Children's Hospital Boston ( Site 0009), Boston, Massachusetts
  - Cincinnati Children's Hospital Medical Center ( Site 0003), Cincinnati, Ohio
  - Children's Hospital of Pittsburgh ( Site 0024), Pittsburgh, Pennsylvania
  - American Research Corporation ( Site 0200), San Antonio, Texas
  - Children's Hospital and Regional Medical Center ( Site 0017), Seattle, Washington
- Germany (3):
  - Medizinische Hochschule Hannover Kinderklinik K10 ( Site 0105), Hanover
  - Klinikum Starnberg ( Site 0107), Starnberg
  - Helios Klinikum Wuppertal GmbH ( Site 0104), Wuppertal
- Poland (3):
  - WSOZ im.T.Browicza w Bydgoszczy ( Site 0800), Bydgoszcz
  - Wojewodzki Specjalistyczny Szpital im. dr W. Bieganskiego w Lodzi ( Site 0810), Lodz
  - MED-POLONIA Sp. z o.o. ( Site 0808), Poznan
- Karolinska Universitetssjukhuset Huddinge. ( Site 0062), Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gonzalez-Peralta RP, Wirth S, Squires RH, Mutschler F, Lang T, Pawlowska M, Sluzewski W, Majda-Stanislawska E, Fischler B, Balistreri WF, Jonas MM, Blondet N, Rosenthal P, Alkhouri N, Romero R, Grandhi A, Castronuovo P, Caro L, Du L, Rosenbloom DIS, Haber BA. Elbasvir/grazoprevir in children aged 3-18 years with chronic HCV genotype 1 or 4 infection: a pharmacokinetic modeling study. Hepatol Commun. 2023 Feb 14;7(3):e0031. doi: 10.1097/HC9.0000000000000031. eCollection 2023 Mar 1. PMID 36790337

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female participants 3 to <18 years of age with chronic hepatitis C virus (HCV) genotype 1 (GT1) or GT4 were enrolled at 14 global study sites.
Groups:
- Age Cohort 1: 12 to <18 Years: Mini and Expanded: Pediatric participants 12 to <18 years of age received elbasvir (EBR) 50 mg / grazoprevir (GZR) 100 mg fixed dose combination (FDC) tablets once daily for 12 weeks.
- Age Cohort 2: 7 to <12 Years: Mini and Expanded: Participants who are 7 to <12 years of age received EBR/GZR 30 mg/60 mg pediatric granules once daily for 12 weeks.
- Age Cohort 3: 3 to <7 Years: Mini: Participants who are 3 to <7 years of age received a pediatric formulation of EBR/GZR (weight-based dosing) once daily for 12 weeks. The Mini cohort consists of the first 7 participants enrolled into Age Cohort 3. Participants <20 kg received EBR/GZR 15 mg/30 mg, and participants ≥20 kg received EBR/GZR 15 mg/50 mg.
- Age Cohort 3: 3 to <7 Years: Expanded: Participants who are 3 to <7 years of age received a pediatric formulation of EBR/GZR 25 mg/50 mg once daily for 12 weeks. The Expanded cohort consists of 11 participants enrolled after the Mini Cohort of 7 participants.
Period: Overall Study
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Started | 22 | 17 | 7 | 11
Completed | 22 | 17 | 7 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Age Cohort 1: 12 to <18 Years: Mini and Expanded: Pediatric participants 12 to <18 years of age received EBR/GZR 50 mg/100 mg FDC tablets once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded | Total
Number analyzed (Participants) | 22 | 17 | 7 | 11 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.1 (1.9) | 8.7 (1.2) | 3.7 (0.8) | 4.8 (1.3) | 9.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 3 | 8 | 29
  Male | 11 | 10 | 4 | 3 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 0 | 6
  Not Hispanic or Latino | 19 | 14 | 6 | 11 | 50
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 17 | 7 | 11 | 56
  More than one race | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Dosing to 24 Hours Postdose (AUC0-24hr) of EBR at Steady State
Description: The AUC0-24hr of EBR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: All randomized and treated participants who complied with the protocol sufficiently to ensure that their pharmacokinetic (PK) data was likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
µM*hr | 2.41 [1.97 to 2.94] | 2.79 [2.31 to 3.37] | 1.71 [1.36 to 2.15] | 3.15 [2.52 to 3.96]

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of EBR
Description: The Cmax of EBR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: All randomized and treated participants who complied with the protocol sufficiently to ensure that their PK data was likely to exhibit the effects of treatment, according to the underlying scientific model, are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
µM | 0.19 [0.15 to 0.23] | 0.21 [0.17 to 0.25] | 0.14 [0.11 to 0.19] | 0.28 [0.22 to 0.36]

3. Primary Outcome: Steady State Predose Drug Concentration (Ctrough) of EBR
Description: The Ctrough of EBR at steady state (Week 4) was determined at steady state prior to dosing in each cohort.
Time Frame: Week 4: Predose
Population: All randomized and treated participants who complied with the protocol sufficiently to ensure that their PK data was likely to exhibit the effects of treatment, according to the underlying scientific model, are included. One participant in Age Cohort 2: 7 to <12 Years: Mini and Expanded had missing Ctrough data.
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 16 | 7 | 11
nM | 59.76 [47.20 to 75.67] | 59.43 [48.67 to 72.58] | 34.61 [28.00 to 42.77] | 68.92 [54.32 to 87.44]

4. Primary Outcome: Apparent Clearance (CL/F) of EBR at Steady State
Description: The CL/F of EBR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
L/hr | 23.53 [19.25 to 28.75] | 12.21 [10.10 to 14.75] | 9.94 [7.89 to 12.53] | 8.98 [7.16 to 11.27]

5. Secondary Outcome: Percentage of Participants With ≥1 Adverse Event (AE)
Description: The percentage of participants with ≥1 AE is reported in each cohort. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 36 weeks
Population: All randomized participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
Percentage of Participants | 81.8 | 76.5 | 85.7 | 81.8

6. Secondary Outcome: Percentage of Participants Discontinuing Study Treatment Due to an AE
Description: The percentage of participants discontinuing study therapy due to an AE is reported in each cohort. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Up to 12 weeks
Population: All randomized participants who received ≥1 dose of study drug are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
Percentage of Participants | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks After Completing Treatment (SVR12)
Description: The percentage of participants achieving SVR12, defined as hepatitis C virus (HCV) ribonucleic acid (RNA) < lower limit of quantification (LLOQ) 12 weeks after completing study therapy, was determined in each cohort.
Time Frame: Week 24
Population: All randomized participants who received ≥1 dose of study treatment are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
Percentage of Participants | 100.0 [84.6 to 100.0] | 100.0 [80.5 to 100.0] | 100.0 [59.0 to 100.0] | 100.0 [71.5 to 100.0]

8. Primary Outcome: AUC0-24hr of GZR at Steady State
Description: The AUC0-24hr of GZR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µM*hr
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
µM*hr | 1.45 [1.08 to 1.94] | 1.42 [1.00 to 2.02] | 0.77 [0.48 to 1.23] | 1.66 [1.16 to 2.39]

9. Primary Outcome: Cmax of GZR
Description: The Cmax of GZR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: µM
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 17 | 7 | 11
µM | 0.25 [0.17 to 0.35] | 0.19 [0.12 to 0.31] | 0.09 [0.05 to 0.18] | 0.29 [0.18 to 0.47]

10. Primary Outcome: Ctrough of GZR
Description: The Ctrough of GZR at steady state (Week 4) was determined at steady state prior to dosing in each cohort.
Time Frame: Week 4: Predose
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: nM
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 22 | 16 | 7 | 11
nM | 16.20 [12.27 to 21.38] | 16.27 [11.97 to 22.10] | 13.79 [9.55 to 19.90] | 16.17 [12.78 to 20.45]

11. Primary Outcome: CL/F of GZR at Steady State
Description: The CL/F of GZR at steady state (Week 4) was determined in each cohort.
Time Frame: Week 4: Predose and 0.5, 1, 2, 3, 4, 6, 8, 10, and 24 hours postdose
Population: No participants are included in the analysis as the CL/F of GZR was not calculable due to nonlinear PK.
Arm/Group | Age Cohort 1: 12 to <18 Years: Mini and Expanded | Age Cohort 2: 7 to <12 Years: Mini and Expanded | Age Cohort 3: 3 to <7 Years: Mini | Age Cohort 3: 3 to <7 Years: Expanded
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 36 weeks for nonserious AEs (NSAEs) and serious AEs (SAEs), and up to approximately 49 weeks for all-cause mortality.
Description: All participants who received ≥1 dose of study drug are included. All-cause mortality is based on all randomized participants.
Groups:
- Age Cohort 1: 12 to < 18 Years: Pediatric participants 12 to <18 years of age received EBR/GZR 50 mg/100 mg FDC tablets once daily for 12 weeks.
- Age Cohort 2: 7 to < 12 Years: Participants who are 7 to <12 years of age received EBR/GZR 30 mg/60 mg pediatric granules once daily for 12 weeks.
- Age Cohort 3 Mini: 3 to < 7 Years: Participants who are 3 to <7 years of age received a pediatric formulation of EBR/GZR (weight-based dosing) once daily for 12 weeks. The Mini cohort consists of the first 7 participants enrolled into Age Cohort 3. Participants <20 kg received EBR/GZR 15 mg/30 mg, and participants ≥20 kg received EBR/GZR 15 mg/50 mg.
- Age Cohort 3 Expanded: 3 to < 7 Years: Participants who are 3 to <7 years of age received a pediatric formulation of EBR/GZR 25 mg/50 mg once daily for 12 weeks. The Expanded cohort consists of 11 participants enrolled after the Mini Cohort of 7 participants.
Arm/Group | Age Cohort 1: 12 to < 18 Years | Age Cohort 2: 7 to < 12 Years | Age Cohort 3 Mini: 3 to < 7 Years | Age Cohort 3 Expanded: 3 to < 7 Years
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/17 | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/22 | 0/17 | 0/7 | 1/11
Other Adverse Events (participants affected / at risk) | 17/22 | 13/17 | 6/7 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort 1: 12 to < 18 Years (N=22) | Age Cohort 2: 7 to < 12 Years (N=17) | Age Cohort 3 Mini: 3 to < 7 Years (N=7) | Age Cohort 3 Expanded: 3 to < 7 Years (N=11)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Age Cohort 1: 12 to < 18 Years (N=22) | Age Cohort 2: 7 to < 12 Years (N=17) | Age Cohort 3 Mini: 3 to < 7 Years (N=7) | Age Cohort 3 Expanded: 3 to < 7 Years (N=11)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 3 (5)
Energy increased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (3)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (7) | 1 (2) | 1 (1) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (4) | 1 (1) | 3 (3)
Rhinitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (3)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (14) | 2 (4) | 0 (0) | 2 (3)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Behaviour disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Provisional tic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study may be published or presented at scientific meetings. The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication of multicenter studies only in their entirety and not as individual site data. If publication activity is not directed by the sponsor, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03379506/Prot_SAP_000.pdf